CLINICAL TRIAL: NCT01925170
Title: Evaluation of Low-dose Molecular Breast Imaging as a Screening Tool in Women With Mammographically Dense Breasts and Increased Risk of Breast Cancer
Brief Title: Low Dose Molecular Breast Imaging as a Screening Tool for Women With Dense Breasts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Deborah Rhodes, Associate Professor of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1337-05 Part B
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-07

CONDITIONS: Breast Cancer
Keywords: Dense breast tissue; Breast Cancer Screening; Molecular Breast Imaging; Breast Cancer; Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Technetium Tc 99m Sestamibi

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mammography and Molecular Breast Imaging (Experimental): Participants underwent conventional mammography and molecular breast imaging after a 740-millibecquerel (mBQ) (8-mCi) Technetium (99mTc) sestamibi injection.
  Interventions: Device: Molecular Breast Imaging; Device: Conventional Mammography; Drug: Technetium (99mTc) sestamibi

INTERVENTIONS:
Device: Molecular Breast Imaging — Molecular breast imaging is a new nuclear medicine technique for imaging the breast. It uses small field of view semiconductor-based gamma cameras that use Cadmium Zinc Telluride detectors. These have superior spatial and energy resolution to conventional sodium iodide detectors.
Device: Conventional Mammography — Mammography is the process of using low-energy X-rays (usually around 30 kVp) to examine the human breast and is used as a diagnostic and a screening tool.
Drug: Technetium (99mTc) sestamibi — Technetium (99mTc) sestamibi is a pharmaceutical agent used in nuclear medicine imaging. The drug is a coordination complex consisting of the radioisotope technetium-99m bound to six methoxyisobutylisonitrile (MIBI) ligands.
  Other Names: Cardiolite

SUMMARY:
A new test for breast cancer screening, molecular breast imaging (MBI) may be more sensitive than mammography for detecting breast cancer in women with dense breasts. The purpose of this study is to see if MBI using a low dose of gamma radiation can find cancers not seen on mammography.

Hypotheses: 1. Low-Dose MBI has a significantly higher sensitivity and specificity and equal or higher positive predictive value than SM in women age 40 and older with mammographically dense breasts. 2. Low-dose MBI has comparable sensitivity and specificity to that previously achieved with MBI using a higher dose of radiation. 3. MBI produces a low false positive rate (specificity >90%) that permits its use as a screening tool in this patient population.

DETAILED DESCRIPTION:
A previous study demonstrated that the addition of MBI using 20 mCi Tc-99m sestamibi to screening mammography (SM) increased diagnostic yield for breast cancer in dense breasts (supplemental yield of 7.5/1000 screened). After implementing radiation dose reduction techniques, the performance of incident SM and prevalent screen MBI in women with dense breasts will be compared.

Methods:

Women presenting for SM with heterogeneously or extremely dense breasts on past prior SM were enrolled and underwent digital SM and MBI. Study information was sent to all eligible patients in advance of their scheduled SM explaining the study and offering them participation. Eligible patients who requested to participate were offered an MBI on the same day as their SM or within 21 days of the SM. Participants may have participated in this screening study up to two times provided at least 24 months had elapsed since the initial MBI scan. This time period was selected as the average time for a tumor to double in size is approximately 20 months. Hence a 24 month time interval between MBI studies was to enable detection of interval cancers or cancers that were too small to be detected in the initial MBI scan.

MBI was performed with 8 mCi Tc-99m sestamibi and dual-head cadmium zinc telluride detectors. SMs were read independently; MBIs were read in comparison with SM. MBIs were assigned an assessment score of 1-5 which parallels BI-RADS; scores of 3-5 on MBI were considered positive.

ELIGIBILITY:
Inclusion Criteria:

* Past prior SM interpreted as negative or benign [Breast Imaging Reporting and Data System (BI-RADS) Category 1 or 2]
* Past prior SM interpreted as heterogeneously dense or extremely dense

Exclusion Criteria:

* Subject is unable to understand and sign the consent form
* Subject is pregnant or lactating
* Subject is physically unable to sit upright and still for 40 minutes
* Subject has self-reported signs or symptoms of breast cancer (palpable mass, bloody nipple discharge, axillary mass, etc.)
* Subject has had needle biopsy within 3 months, or breast surgery within 1 year prior to the study
* Subject is currently taking tamoxifen, Evista (raloxifene), Zoladex or an aromatase inhibitor for adjuvant therapy or chemoprevention.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1638 (Actual)
Dates: Start 2009-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J Rhodes, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Rhodes DJ, Hruska CB, Phillips SW, Whaley DH, O'Connor MK. Dedicated dual-head gamma imaging for breast cancer screening in women with mammographically dense breasts. Radiology. 2011 Jan;258(1):106-18. doi: 10.1148/radiol.10100625. Epub 2010 Nov 2. PMID 21045179
- See also: 1337-05 Part A, High-Dose Molecular Breast Imaging — http://clinicaltrials.gov/show/NCT00620373

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women for the Part B low dose study were enrolled between 5/11/2009 and 3/8/2012.
Period: Overall Study
Arm/Group | Mammography and Molecular Breast Imaging
Started | 1638
Completed | 1585
Not Completed | 53
Not completed — Unverified cancer status | 53

BASELINE CHARACTERISTICS:
Arm/Group | Mammography and Molecular Breast Imaging
Number analyzed (Participants) | 1638
Age, Continuous [Mean (Full Range); unit: years] — At the beginning of the study, the protocol inclusion criteria allowed women aged 25 years and older to participate. Between the dates of 5/11/09 and 4/20/10 there were 13 women under age 40 enrolled. On 4/20/2010 a protocol revision was approved by the Institutional Review Board to allow women aged 40 and older. In the final analyzable dataset of 1585 women who completed the study and had reference standard, 6 women were under age 40.
  years | 58.1 [31 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1638
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 1605
  More than one race | 0
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 1638
Menopausal Status [Number; unit: participants]
  Premenopausal | 355
  Peri-menopausal | 186
  Postmenopausal | 1021
  Surgical Menopause | 76
Mammographic Breast Density [Number; unit: participants] — Eligibility was determined by density assessed on a previous mammogram prior to study entry; mammographic density reported refers to density assessed from the study mammogram.
  participants
    Almost entirely fat | 0
    Scattered fibroglandular densities | 149
    Heterogeneously dense | 1259
    Extremely dense | 230
Risk Factors [Number; unit: participants] — Although participants may have qualified for multiple risk factor categories, they were assigned to only one risk factor category in this table. These risk factors are listed in order of priority. The last two risk factors with respect to first and second-degree relatives with a history of breast cancer refer to subjects who qualified on the basis of family history but did not meet the Gail or Claus model risk threshold levels.
  The Gail risk model focuses on nongenetic risk factors, with limited information on family history. The Claus risk model focuses on genetic risk factors.
  participants
    Known mutation in BRCA1 or BRCA2 genes | 3
    Chest, mediastinal, or axillary irradiation | 5
    Personal history of breast cancer | 166
    Prior biopsy showing hyperplasia, etc. | 21
    Gail or Claus model lifetime risk ≥ 20% | 78
    Gail model 5 year risk ≥ 2.5% | 203
    Gail model 5 year risk ≥ 1.7% | 360
    1 first-deg relative with history of breast cancer | 53
    2 2nd-deg relatives with history of breast cancer | 56
    None of the above risk factors | 693
Mammogram Prior to Study Entry [Number; unit: participants] — A total of 7 women under the age of 50 with no prior mammogram were enrolled.
  participants
    < 425 days | 1310
    425-730 days | 301
    >730 days | 20
    None | 7
Molecular Breast Imaging Prior to Study Entry [Number; unit: participants]
  < 425 days | 0
  415- 730 days | 8
  > 730 days | 171
  None | 1459
Breast Density of Participants with No Prior Mammogram [Number; unit: participants]
  Scattered fibroglandular densities | 2
  Heterogeneously dense breasts | 5
  Participants with Prior Mammogram | 1631

OUTCOME MEASURES:

1. Primary Outcome: Cancer Detection Rate Per 1000 Women Screened, by Breast Density
Description: The cancer detection rate per 1000 women screened is the estimate of the number of women with positive results from a screening test.
Time Frame: Within 21 days of mammography
Measure: Number (95% Confidence Interval); unit: cancers per 1000 women screened
Groups:
- Mammography Only: For this reporting arm, the interpretation and analysis was done with mammography only.
- Mammography With Adjunct MBI: For this reporting arm, the interpretation and analysis was done with both mammography and MBI together.
- Molecular Breast Imaging Alone: For this reporting arm, the interpretation and analysis was done with gamma imaging only.
Arm/Group | Mammography Only | Mammography With Adjunct MBI | Molecular Breast Imaging Alone
Number analyzed (Participants) | 1585 | 1585 | 1585
cancers per 1000 women screened
  All densities | 3.2 [1.3 to 7.4] | 12.0 [7.7 to 18.6] | 10.7 [6.7 to 17.1]
  Scattered fibroglandular densities | 0 [0 to 26.2] | 21.0 [7.2 to 59.9] | 21.0 [7.2 to 59.9]
  Heterogeneously dense | 3.3 [1.3 to 8.4] | 10.6 [6.2 to 18.1] | 9.0 [5.0 to 16.0]
  Extremely dense | 4.5 [0.2 to 25.2] | 13.6 [4.6 to 39.1] | 13.6 [4.6 to 39.1]
Statistical Analysis 1: Comparison: Mammography Only vs Mammography With Adjunct MBI; Comparison of the two groups for all densities, significant difference p ≤ 0.05; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Mammography Only vs Molecular Breast Imaging Alone; Comparison of two groups for all densities; significant difference p ≤ 0.05; Test type: Superiority or Other; p = 0.004, t-test, 2 sided

2. Secondary Outcome: Specificity
Description: Specificity measures the percentage of negatives which are correctly identified as such.
Time Frame: Within 21 days of mammography
Population: The analysis population only included participants with a verified negative cancer status at 12 months after the initial screening (mammography and MBI).
Measure: Number (95% Confidence Interval); unit: percentage of true negatives
Arm/Group | Mammography Only | Mammography With Adjunct MBI | Molecular Breast Imaging Alone
Number analyzed (Participants) | 1564 | 1564 | 1564
percentage of true negatives | 89.1 [87.5 to 90.6] | 83.4 [81.4 to 85.1] | 93.5 [92.1 to 94.6]
Statistical Analysis 1: Comparison: Mammography Only vs Mammography With Adjunct MBI; Significant difference p ≤ 0.05; Test type: Superiority or Other; p < 0.001, McNemar
Statistical Analysis 2: Comparison: Mammography Only vs Molecular Breast Imaging Alone; Significant difference p ≤ 0.05; Test type: Superiority or Other; p < 0.0001, McNemar

3. Secondary Outcome: Sensitivity for All Cancers Diagnosed
Description: Sensitivity measures the percentage of actual positives which are correctly identified as such.
Time Frame: Within 21 days of mammography
Population: The analysis population only included participants with a verified cancer status at 12 months after the initial screening. 21 participants out of the total study population of 1585 were diagnosed with cancer.
Measure: Number (95% Confidence Interval); unit: percentage of actual positives
Arm/Group | Mammography Only | Mammography With Adjunct MBI | Molecular Breast Imaging Alone
Number analyzed (Participants) | 21 | 21 | 21
percentage of actual positives | 23.8 [10.6 to 45.1] | 90.5 [71.1 to 97.3] | 81.0 [60.0 to 91.3]
Statistical Analysis 1: Comparison: Mammography Only vs Mammography With Adjunct MBI; Significant difference p ≤ 0.05; Test type: Superiority or Other; p < 0.001, McNemar
Statistical Analysis 2: Comparison: Mammography Only vs Molecular Breast Imaging Alone; Significant difference p ≤ 0.05; Test type: Superiority or Other; p = 0.004, McNemar

4. Secondary Outcome: Recall Rate
Description: Recall rate was defined as the percentage of participants recalled for follow-up studies initiated because of abnormal findings with mammography or MBI.
Time Frame: 12 months after mammography and MBI
Population: The analysis population only included participants with a verified cancer status at 12 months after the initial screening (mammography and MBI).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mammography Only | Mammography With Adjunct MBI | Molecular Breast Imaging Alone
Number analyzed (Participants) | 1585 | 1585 | 1585
percentage of participants | 11.0 [9.6 to 12.7] | 17.6 [15.8 to 19.6] | 7.5 [6.3 to 8.9]
Statistical Analysis 1: Comparison: Mammography Only vs Mammography With Adjunct MBI; Significant difference p ≤ 0.05; Test type: Superiority or Other; p < 0.001, McNemar
Statistical Analysis 2: Comparison: Mammography Only vs Molecular Breast Imaging Alone; Significant difference p ≤ 0.05; Test type: Superiority or Other; p < 0.001, McNemar

5. Secondary Outcome: Biopsy Rate
Description: Biopsy rate = number of participants who had a biopsy/number of number of participants analyzed.
Time Frame: 12 months after mammography and MBI
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mammography Only | Mammography With Adjunct MBI | Molecular Breast Imaging Alone
Number analyzed (Participants) | 1585 | 1585 | 1585
percentage of participants | 1.3 [0.8 to 1.9] | 4.2 [3.3 to 5.3] | 3.2 [2.5 to 4.2]
Statistical Analysis 1: Comparison: Mammography Only vs Mammography With Adjunct MBI; Significant difference p ≤ 0.05; Test type: Superiority or Other; p < 0.001, McNemar
Statistical Analysis 2: Comparison: Mammography Only vs Molecular Breast Imaging Alone; Significant difference p ≤ 0.05; Test type: Superiority or Other; p < 0.001, McNemar

ADVERSE EVENTS:
Time Frame: Participants were followed for adverse events while they were on the study.
Arm/Group | Mammography and Molecular Breast Imaging
Serious Adverse Events (participants affected / at risk) | 0/1585
Other Adverse Events (participants affected / at risk) | 0/1585

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No